CLINICAL TRIAL: NCT05415111
Title: The Adjunctive Effect of Soft Tissue Augmentation Procedures on the Surgical Treatment of Moderate-severe Peri-implantitis: A Randomized Controlled Clinical Trial.
Brief Title: The Adjunctive Effect of Soft Tissue Augmentation Procedures of Moderate-severe Peri-implantitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadja Naenni (Other)
Responsible Party: Sponsor-Investigator, Nadja Naenni, PD Dr. med. dent, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022 - 462
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Peri-Implantitis
Keywords: tissue augmentation of moderate-severe peri-implantitis; implantoplasty; collagen matrix; autogenous connective tissue graft
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Study specific intervention is the placement of a soft tissue autogenous graft (SCTG) or soft tissue substitute (VCMX) in addition to bone grafting of periimplantitis-affected implants. Study specific control intervention is the placement of a bone graft at periimplantitis-affected implants. No soft tissue grafts will be placed. The bone graft will remain permanently in the patients.
Masking Description: Masking is not possible for the intended interventions, as the harvest of the SCTG requires an additional surgical site at the palate, which will be recognized by the patient. The investigators will also be aware of the type of procedure, as both follow different operation procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subepithelial connective tissue group (SCTG) (Active Comparator): A SCTG will be harvested from the patient's palate with a dimension dependent on the size of the peri-implant osseous defect. The technique of harvesting a soft tissue grafting is well described and established in the literature. Following the administration of local anesthesia, the SCTG will be harvested using a single incision technique. The periosteum will be left intact. The thickness of the SCTG will be at least 1.5mm. A cross suture will be used to close the palatal incision.
  The SCTG will be placed on the buccal exposed implant threads (above the DBBM-C) exceeding 1mm in a coronal and apical direction, 3mm in a mesial and distal direction and then immobilized using a horizontal mattress connecting it to the lingual or palatal flap. The flaps are then closed primarily and tension-free following a horizontal periosteal releasing incision.
  Interventions: Procedure: Subepithelial connective tissue
- Volume stable Collagen Matrix group (VCMX) (Active Comparator): A VMCX (FibroGide®) will be hydrated in sterile saline, trimmed and adjusted to a dimension dependent on the size of the osseous peri-implant defect. The VCMX will then be placed as described above and then immobilized using a horizontal mattress connecting it to the lingual or palatal flap. The flaps are then closed primarily and tension-free following a horizontal periosteal releasing incision.
  Interventions: Procedure: Volume stable Collagen Matrix
- No soft tissue augmentation (GBR) (Sham Comparator): No barrier membranes will be placed. After filling the defect with the bone substitute, the flaps are closed primarily and tension-free following a horizontal periosteal releasing incision.
  Interventions: Procedure: No soft tissue augmentation

INTERVENTIONS:
Procedure: Subepithelial connective tissue — Study specific intervention is the placement of a soft tissue autogenous graft (SCTG) in addition to bone grafting of periimplantitis-affected implants.
  Arms: Subepithelial connective tissue group (SCTG)
Procedure: Volume stable Collagen Matrix — Study specific intervention is the placement of a soft tissue substitute (VCMX) in addition to bone grafting of periimplantitis-affected implants.
  Arms: Volume stable Collagen Matrix group (VCMX)
Procedure: No soft tissue augmentation — Study specific control intervention is the placement of a bone graft at periimplantitis-affected implants. No soft tissue grafts will be placed.
  Arms: No soft tissue augmentation (GBR)

SUMMARY:
The key objective of the study is to compare the effects of soft tissue augmentation using a volume stable collagen matrix or autogenous connective tissue graft or no soft tissue augmentation in addition to bone grafting/implantoplasty in patients who undergo surgical therapy of peri-implantitis with respect to clinical resolution of the infection.

DETAILED DESCRIPTION:
The global burden of periimplantitis is expected to rise with the increasing popularity of dental implants as a replacement option. While many therapeutic interventions have been proposed, none have been proven superior. Surgical therapy is often indicated to gain access to the plaque infected implant threads and bone defects. Implantoplasty of suprabony defects have shown good results although adverse effects like soft tissue recession are common.

Thin mucosa results in compromised outcomes following various surgical interventions around implants with increased recession and aesthetic failures. It has also been associated with increased marginal bone loss and severity of periimplantitis. Application of autogenous connective tissue grafts during surgical therapy of periimplantitis to increase the keratinised mucosa widths or attenuate post-implantoplasty recession showed promising results.

No randomized controlled clinical trials investigating the effects of additional soft tissue augmentation with implantoplasty on periimplantitis lesions have been done so far. In addition, few have evaluated patient reported outcome measures, included non-European subjects and none reported on soft tissue alterations. The effect of soft tissue substitutes on surgical periimplantitis therapy remains unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old (UZH, FRA) or > 21 years old (SIN), male and female.
2. Diagnosed with periimplantitis of at least 1 implant in function for at least 1 year Diagnostic criteria

   * Presence of bleeding and/or suppuration on gentle probing.
   * Probing depths of ≥6 mm.
   * Bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant.
3. Periodontal health (including previously treated periodontitis patients with reduced but healthy periodontium)
4. Good oral hygiene (full mouth plaque score <25%)
5. Adequate control of inflammation (full mouth BOP <25%)
6. Signed informed consent form

Exclusion Criteria:

1. Pregnant or lactating female patient at inclusion
2. Allergy or objection to porcine and bovine implantable biomaterials
3. Allergy to Penicillin or NSAIDs
4. Known or suspected non-compliance, drug or alcohol abuse
5. Inability to follow the procedures of the study, e.g. due to language/ comprehension problems, psychological disorders, dementia, etc. of the participant
6. Smoking > 15 cigarettes a day
7. Active periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Absence of bleeding/ suppuration on probing | 6 months after surgery
  A parameter for monitoring periodontal conditions
Increase in probing depth ≤ 1mm | 6 months after surgery
  A parameter for monitoring periodontal conditions
Absence of additional bone loss after therapy of more than 5mm from radiographic baseline | 6 months after surgery
  A parameter for monitoring periodontal conditions

SECONDARY OUTCOMES:
Profilometric changes around the treated implant | 6 months after surgery
  The profilometric changes will be evaluated based on intra-oral scans
Profilometric changes around the treated implant | 1 year after surgery
  The profilometric changes will be evaluated based on intra-oral scans
Profilometric changes around the treated implant | 3 year after surgery
  The profilometric changes will be evaluated based on intra-oral scans
Profilometric changes around the treated implant | 5 year after surgery
  The profilometric changes will be evaluated based on intra-oral scans
Early wound healing | 1 month after surgery
  The index assesses wound healing using scores from 1 to 5: a wound with very poor healing receives a score of 1, whereas excellent healing receives a score of 5
Early wound healing | 2 month after surgery
  The index assesses wound healing using scores from 1 to 5: a wound with very poor healing receives a score of 1, whereas excellent healing receives a score of 5
Radiographic evaluation of the amount of hard tissue | 6 months after surgery
  evaluation of the marginal bone level changes
Radiographic evaluation of the amount of hard tissue | 1 year after surgery
  evaluation of the marginal bone level changes
Radiographic evaluation of the amount of hard tissue | 3 years after surgery
  evaluation of the marginal bone level changes
Radiographic evaluation of the amount of hard tissue | 5 years after surgery
  evaluation of the marginal bone level changes
Oral Health Impact Profile-14 | 6 months after surgery
  Patient's questionnaire - has 14 items with answers rated on a 5-point Likert scale (from 1 = never to 5 = very often) to indicate a level of different problems related to oral health
Oral Health Impact Profile-14 | 1 year after surgery
  Patient's questionnaire - 14 items with answers rated on a 5-point Likert scale (from 1 = never to 5 = very often) to indicate a level of different problems related to oral health
Oral Health Impact Profile-14 | 3 years after surgery
  Patient's questionnaire - has 14 items with answers rated on a 5-point Likert scale (from 1 = never to 5 = very often) to indicate a level of different problems related to oral health
Oral Health Impact Profile-14 | 5 years after surgery
  Patient's questionnaire - has 14 items with answers rated on a 5-point Likert scale (from 1 = never to 5 = very often) to indicate a level of different problems related to oral health

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Naenni, Dr., Principal Investigator — University of Zurich
Locations (3):
- Department of Oral Surgery and Implantology, Centre for Dentistry and Oral Medicine (Carolinum), Johann Wolfgang Goethe-University Frankfurt, Frankfurt, Germany
- National Dental Centre Singapore, Singapore, Singapore
- Clinic of Reconstructive Dentistry, Center of Dental Medicine University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No